CLINICAL TRIAL: NCT02180945
Title: ONYX Evaluation in the Endovascular Treatment of Intracranial Dural Arteriovenous Fistulae. A French, Observational, Prospective, Multicentric, Single Arm and Open Study
Brief Title: ONYX Evaluation in the Endovascular Treatment of Intracranial Dural Arteriovenous Fistulae
Acronym: dAVF
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-ONY-001
Record Dates: First submitted 2014-04-25; First posted 2014-07-03 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Arteriovenous Fistula
Keywords: dAVF; Arteriovenous fistula; ONYX
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intracranial Dural Arteriovenous Fistula: Adult patients requiring endovascular treatment of Intracranial Dural Arteriovenous Fistulae.

SUMMARY:
The objective of this study is to evaluate the safety and performance post last embolization with Onyx

ELIGIBILITY:
Inclusion Criteria:

* The patient has an intracranial dAVF which could be treated by ONYX embolization, whether or not associated to other embolization products.
* The patient is at least 18 years of age.

Exclusion Criteria:

* The patient needs to be treated for the dAVF with another treatment option (for example by surgery) than embolization within a period of less than 6 months (to be counted as from the first treatment)
* The patient participates to another clinical study during the treatment period for his/her dAVF, evaluating another medical devices, procedure or medication.
* The patient refuses to give consent to the collection and processing of data required for centralized monitoring.
* A condition which could jeopardize follow-up of the patient.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the participating centers for whom an intracranial dAVF (not previosly treated) needs to be treated (unrelated to the planned treatment) and who agree to the collection and transmission of related data.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Neurological clinical evolution | 1Month post procedure
  Improved, Stable, Worsened, death
Healing rate | 3-6 months post procedure
  Number of patients with No residual early venous return

SECONDARY OUTCOMES:
Adverse event | 3-6 months after procedure
  The number of adverse events (causing death or otherwise)
Quality of life EQ-5D | pre-procedure and at 3-6 months
  Health State Score increase
Describe functional independence | 1 and 12 months after procedure
  Describe mRS scores assessed by a certified physician
Technical performance of the product | 12 months after procedure
  Volume injected per embolization session

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Cognard, Prof. Dr., Principal Investigator — University Hospital, Toulouse; Frédéric Ricolfi, Prof. Dr., Principal Investigator — Centre Hospitalier Universitaire Dijon; Patrick Courthéoux, Prof. Dr., Principal Investigator — University Hospital, Caen; Laurent Spelle, Prof. Dr., Principal Investigator — Hôpital Beaujon
Locations (1):
- Covidien, Paris, France